CLINICAL TRIAL: NCT02743936
Title: Analysis of Face Mask Leak With Nasal Cannula in Noninvasive Positive Pressure Ventilation: A Randomized Crossover Trial
Brief Title: Mask Leak With Nasal Cannula in Noninvasive Positive Pressure Ventilation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael D. April, Assistant Program Director for Research, Brooke Army Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C.2016.030d
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-08

CONDITIONS: Mechanical Ventilation Pressure High
MeSH Terms: interventions — Cannula

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIPPV with nasal cannula (Experimental): Non-invasive positive pressure ventilation with nasal cannula in place
  Interventions: Device: Nasal cannula; Device: Non-invasive positive pressure ventilation
- NIPPV without nasal cannula (Active Comparator): Non-invasive positive pressure ventilation without nasal cannula
  Interventions: Device: Non-invasive positive pressure ventilation

INTERVENTIONS:
Device: Nasal cannula — Placement of nasal cannula under non-invasive positive pressure ventilation mask
  Other Names: NC
  Arms: NIPPV with nasal cannula
Device: Non-invasive positive pressure ventilation — Non-invasive positive pressure ventilation
  Other Names: NIPPV

SUMMARY:
This is a prospective randomized cross over study of healthy volunteers undergoing continuous positive airway pressure ventilation via a noninvasive ventilation (NIV) mask with and without the addition of nasal cannulas. Mask leak will be measured by the ventilator after 60 seconds of spontaneous resting ventilation, with each subject serving as his or her own control.

DETAILED DESCRIPTION:
This is a randomized cross over study. A convenience sample of staff and resident physicians and physician assistants from the San Antonio Military Medical Center (SAMMC) Department of Emergency Medicine will be used to assess NIPPV mask seal during CPAP administration with and without nasal cannula. Volunteers will be solicited via Grand Rounds and staff meetings at San Antonio Military Medical Center. Subjects will undergo permuted block randomization by random number generator to the order of intervention, mask alone or mask with nasal cannula at 15L/min of oxygen. An emergency medicine trained physician will place equipment and operate the ventilator. After placement of the NIPPV mask and prior to each study intervention period, appropriate adjustments to enhance mask seal will be made as would happen in a therapeutic setting and the volunteer will be allowed up to two minutes to acclimate to continuous noninvasive positive pressure ventilation. Mask leak will be measured by the ventilator unit and will be recorded after 60 seconds of spontaneous restful ventilation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Volunteer for study

Exclusion Criteria:

* Known cardiac disease
* Known pulmonary disease (to include respiratory infections)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D April, MD, PhD, MSc, Principal Investigator — Brooke Army Medical Center
Locations (1):
- San Antonio Military Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Background] Baillard C, Fosse JP, Sebbane M, Chanques G, Vincent F, Courouble P, Cohen Y, Eledjam JJ, Adnet F, Jaber S. Noninvasive ventilation improves preoxygenation before intubation of hypoxic patients. Am J Respir Crit Care Med. 2006 Jul 15;174(2):171-7. doi: 10.1164/rccm.200509-1507OC. Epub 2006 Apr 20. PMID 16627862
- [Background] Ramachandran SK, Cosnowski A, Shanks A, Turner CR. Apneic oxygenation during prolonged laryngoscopy in obese patients: a randomized, controlled trial of nasal oxygen administration. J Clin Anesth. 2010 May;22(3):164-8. doi: 10.1016/j.jclinane.2009.05.006. PMID 20400000
- [Background] Lawes EG, Campbell I, Mercer D. Inflation pressure, gastric insufflation and rapid sequence induction. Br J Anaesth. 1987 Mar;59(3):315-8. doi: 10.1093/bja/59.3.315. PMID 3828180

RESULTS

PARTICIPANT FLOW:
Groups:
- NIPPV With Nasal Cannula First: Non-invasive positive pressure ventilation (NIPPV) with nasal cannula in place followed by NIPPV without nasal cannula in place.
  Nasal cannula: Placement of nasal cannula under non-invasive positive pressure ventilation mask
  Non-invasive positive pressure ventilation: Non-invasive positive pressure ventilation
- NIPPV Without Nasal Cannula First: Non-invasive positive pressure ventilation (NIPPV) without nasal cannula first then NIPPV with nasal cannula
  Nasal cannula: Placement of nasal cannula under non-invasive positive pressure ventilation mask
  Non-invasive positive pressure ventilation: Non-invasive positive pressure ventilation
Period: Overall Study
Arm/Group | NIPPV With Nasal Cannula First | NIPPV Without Nasal Cannula First
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIPPV With Nasal Cannula First | NIPPV Without Nasal Cannula First | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [28 to 36] | 32 [28 to 34] | 31 [28 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Face Mask Leak Measured in Liters Per Minute by the Noninvasive Positive Pressure Ventilation Machine
Description: Face mask leak as measured in liters per minute by the noninvasive positive pressure ventilation machine
Time Frame: 2 minutes after mask placement
Measure: Median (Inter-Quartile Range); unit: Liters per minute
Arm/Group | NIPPV With Nasal Cannula | NIPPV Without Nasal Cannula
Number analyzed (Participants) | 64 | 64
Liters per minute | 0 [0 to 3.3] | 0 [0 to 0.9]

2. Secondary Outcome: Patient Discomfort (Verbal Numerical Rating Scale)
Description: Discomfort scored on a 0-10 verbal numerical rating scale (0 = no discomfort, 10 = most discomfort imaginable)
Time Frame: After study completion (approximately 2 minutes after study start)
Measure: Median (Inter-Quartile Range); unit: Scores on verbal numerical rating scale
Arm/Group | NIPPV With Nasal Cannula | NIPPV Without Nasal Cannula
Number analyzed (Participants) | 64 | 64
Scores on verbal numerical rating scale | 3 [2 to 5] | 1 [1 to 2]

ADVERSE EVENTS:
Arm/Group | NIPPV With Nasal Cannula First | NIPPV Without Nasal Cannula First
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No